CLINICAL TRIAL: NCT01078116
Title: Cost Utility Analyses of Adalimumab Treatment in Patients With Rheumatoid Arthritis
Brief Title: Cost Utility Analyses of Adalimumab Treatment in Patients With Rheumatoid Arthritis (RA)
Acronym: HEOR
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Institute of Political Economical & Social Researches, Greece (Unknown)
Responsible Party: Tina Antachopoulou / Medical Director, Abbott Laboratories Hellas S.A.
Other Study IDs: P10-159
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Adalimumab treatment; Evaluation of the patients' Health Related Quality of Life; Cost of the disease management
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Rheumatoid Arthritis: Eligible rheumatoid arthritis patients treated with adalimumab according to the approved Summary of Product Characteristics (SmPC) in European Union

SUMMARY:
Evaluation of Health Related Quality of Life (HRQL) is of a paramount importance in assessing the impact of rheumatoid arthritis on patients' health status, however when costs associated with rheumatoid arthritis are also taken into account, the information provided may lead to a more balanced view in analyzing the treatment of the disease.

In accordance with the above, the main objective this study was to evaluate the impact of adalimumab treatment not only on patients' Health Related Quality of Life but also on the cost of the disease management. In order to accomplish this the study has been focused on:

1. Estimating the direct and indirect cost incurred by adalimumab treatment.
2. Measuring the Health Related Quality of Life of rheumatoid arthritis patients under adalimumab treatment.
3. Exploring the cost-utility relationship of rheumatoid arthritis patients treated with adalimumab by combining the Health Related Quality of Life of rheumatoid arthritis patients and direct as well as indirect costs due to RA.

More specifically, data related to patients' Health Related Quality of Life and cost associated with rheumatoid arthritis will be recorded for one-year period, and collected at four subsequent visits: baseline, month 3, 6 and 12. The visit before starting treatment with adalimumab will be considered as baseline. This information was used to compare Health Related Quality of Life and cost data before and after adalimumab initiation and therefore identify the effect of adalimumab treatment in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Data concerning patients' Health Related Quality of Life as well as the cost of the disease treatment were collected at four subsequent periods and specifically at baseline (Visit 1), and at months 3, 6 and 12.

Moreover, at baseline patients' socioeconomic, and history of illness data as well as the use of other prescribed medication and costs due to rheumatoid arthritis have been recorded, in order to identify patients' health state before adalimumab treatment initiation.

Patients discontinuing therapy (drop-outs) either due to adverse events or on their own initiative were categorized and analyzed separately, while reasons leading to discontinuation were recorded. Adverse events were not collected in this study with the exception of adverse events leading to withdrawal.

In order to evaluate the cost-utility of adalimumab both the cost of the disease treatment and the Health Related Quality of Life of rheumatoid arthritis patients have been taken into account. The process is described below:

Face-to-face interviews were conducted by the physicians/investigators in charge in all four subsequent periods as well as before adalimumab treatment initiation. A questionnaire, divided into the following sections, was administered: 1. Patients' Sociodemographic Characteristics 2. Measurement of Health Related Quality of Life in Rheumatoid Arthritis patients 3. Cost Assessment

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate or severe active rheumatoid arthritis, who have been prescribed and are receiving adalimumab under normal clinical practice for at least one month and according to the approved Summary of Product Characteristics (SmPC) in the European Union.
* Patients must be willing to consent to data being collected and provided to Abbott Laboratories.

Exclusion Criteria:

* Contraindications according to the SmPC
* Patients should not participate in other observational Abbott study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis, from hospital centres and private physicians, who were prescribed adalimimab according to the approved SmPC in the European Union, prior to the study enrollment
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2007-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thanasis Floros, MD, Study Chair — Abbott Laboratories Hellas S.A.
Locations (10):
- Greece (10):
  - Site Reference ID/Investigator# 32052, Athens
  - Site Reference ID/Investigator# 32068, Athens
  - Site Reference ID/Investigator# 32069, Athens
  - Site Reference ID/Investigator# 32071, Crete
  - Site Reference ID/Investigator# 32072, Ioannina
  - Site Reference ID/Investigator# 32073, Larissa
  - Site Reference ID/Investigator# 32064, Thessaloniki
  - Site Reference ID/Investigator# 32065, Thessaloniki
  - Site Reference ID/Investigator# 32066, Thessaloniki
  - Site Reference ID/Investigator# 32067, Thessaloniki

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab Treatment: Male or female participants with moderate to severe active rheumatoid arthritis treated with adalimumab according to the approved Summary of Product Characteristics (SmPC) in European Union
Period: Overall Study
Arm/Group | Adalimumab Treatment
Started | 124 (121 participants were included in analysis (3 were excluded due to missing case report form data).)
Completed | 76
Not Completed | 48
Not completed — Lost to Follow-up | 17
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 8
Not completed — Lack of effectiveness | 15
Not completed — Case report form not completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab Treatment
Number analyzed (Participants) | 121
Age Continuous [Mean (Standard Deviation); unit: years] — Based on population of 121 participants analyzed.
  years | 56.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Based on population of 121 participants analyzed.
  Participants
    Female | 100
    Male | 21
Region of Enrollment [Number; unit: participants] — Based on population of 121 participants analyzed.
  participants
    Greece | 121

OUTCOME MEASURES:

1. Primary Outcome: Estimation of the Direct and Indirect Cost Incurred by Adalimumab Treatment
Description: Direct and indirect per-participant costs were estimated at Baseline (enrollment visit) for the 3-month period prior to initiation of adalimumab treatment, and at 3, 6 and 12 months following initiation of treatment. Direct costs included pharmaceutical costs, diagnostic and monitoring test costs, hospitalization costs, rheumatologist's costs, social insurance rheumatologist's costs, other specialists costs, physiotherapy costs, rehabilitation cost, home care cost, equipment cost and transportation cost. Indirect costs refer to loss of income due to rheumatoid arthritis disability.
Time Frame: Enrollment visit (Baseline), month 3, month 6, month 12
Population: Analysis is based on the number of participants completing the assessments at each visit.
Measure: Mean (Standard Deviation); unit: Euros
Arm/Group | Adalimumab Treatment
Number analyzed (Participants) | 121
Euros
  Direct Costs at Baseline (n=121) | 272.99 (383.48)
  Indirect Costs at Baseline (n=13) | 1162.62 (1146.60)
  Direct Costs at 3 months (n=104) | 2662.73 (446.86)
  Indirect Costs at 3 months (n=8) | 659.13 (648.82)
  Direct Costs at 6 months (n=91) | 2692.28 (243.82)
  Indirect Costs at 6 months (n=4) | 500.00 (336.65)
  Direct Costs at 12 months (n=76) | 2649.42 (533.47)
  Indirect Costs at 12 months (n=1) | 580.00 (0)

2. Primary Outcome: Health Related Quality of Life (European Quality of Life 5 Dimensions)
Description: European Quality of Life 5 Dimensions (EQ-5D) is a generic health related quality of life instrument which assesses 5 health dimensions on a scale of 1 (no problems) to 5 (worst health). An overall score is derived ranging from -.59 to +1; a higher score indicates better health.
Time Frame: Enrollment visit (Baseline), month 3, month 6, month 12
Population: Analysis is based on the number of participants completing the assessments at each visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Adalimumab Treatment
Number analyzed (Participants) | 121
Units on a scale
  EQ-5D Score at Baseline | 0.43 (0.16)
  EQ-5D Score at 3 months | 0.53 (0.23)
  EQ-5D Score at 6 months | 0.56 (0.23)
  ED-5D Score at 12 months | 0.62 (0.25)

3. Primary Outcome: Health Related Quality of Life (Health Assessment Questionnaire)
Description: Health Assessment Questionnaire (HAQ) is designed to assess patients' abilities to perform activities of daily living. Scores range between 0 and 3, where higher values represent worse outcomes.
Time Frame: Enrollment visit (Baseline), month 3, month 6, month 12
Population: Analysis is based on the number of participants completing the assessment at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab Treatment
Number analyzed (Participants) | 121
units on a scale
  HAQ Score at Baseline | 1.33 (0.70)
  HAQ Score at 3 months | 0.95 (0.80)
  HAQ Score at 6 months | 0.83 (0.64)
  HAQ Score at 12 months | 0.62 (0.64)

4. Primary Outcome: Health Related Quality of Life (Medical Outcome Study Short Form 36)
Description: Medical Outcome Study Short Form 36 (MOS SF-36) is a generic health related quality of life assessment that consists of 36 questions within 8 domains. Results from each domain are summarized and transformed into a scale ranging from 0 (worst) to 100 (best).
Time Frame: Enrollment visit (Baseline), month 3, month 6, month 12
Population: Analysis is based on the number of participants completing the assessment at each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Adalimumab Treatment
Number analyzed (Participants) | 121
Units on a scale
  Physical Functioning Score at Baseline | 33.5 (26.0)
  Physical Functioning Score at 3 months | 50.0 (29.4)
  Physical Functioning Score at 6 months | 56.4 (27.8)
  Physical Functioning Score at 12 months | 60.0 (28.9)
  Role Physical Score at Baseline | 18.7 (34.0)
  Role Physical Score at 3 months | 36.8 (43.3)
  Role Physical Score at 6 months | 41.0 (43.7)
  Role Physical Score at 12 months | 51.0 (45.0)
  Bodily Pain Score at Baseline | 37.2 (20.6)
  Bodily Pain Score at 3 months | 55.5 (23.5)
  Bodily Pain Score at 6 months | 60.0 (24.5)
  Bodily Pain Score at 12 months | 63.2 (23.1)
  General Health Score at Baseline | 33.8 (20.5)
  General Health Score at 3 months | 45.4 (23.5)
  General Health Score at 6 months | 48.5 (23.5)
  General Health Score at 12 months | 52.8 (23.1)
  Vitality Score at Baseline | 35.8 (20.2)
  Vitality Score at 3 months | 48.7 (21.0)
  Vitality Score at 6 months | 51.0 (19.6)
  Vitality Score at 12 months | 56.2 (18.4)
  Social Functioning Score at Baseline | 47.4 (33.5)
  Social Functioning Score at 3 months | 61.5 (28.5)
  Social Functioning Score at 6 months | 63.7 (29.5)
  Social Functioning Score at 12 months | 70.5 (26.3)
  Role Emotional Score at Baseline | 32.0 (44.0)
  Role Emotional Score at 3 months | 50.7 (47.4)
  Role Emotional Score at 6 months | 54.6 (47.5)
  Role Emotional Score at 12 months | 70.2 (42.1)
  Mental Health Score at Baseline | 48.0 (21.0)
  Mental Health Score at 3 months | 57.1 (20.0)
  Mental Health Score at 6 months | 58.5 (20.0)
  Mental Health Score at 12 months | 61.4 (16.8)

5. Primary Outcome: Cost-Utility Relationship of Rheumatoid Arthritis Patients Treated With Adalimumab Using Incremental Cost-Effectiveness Approach (ICER)
Description: The ICER calculation is based on comparison of differences in costs and utilities (based on Quality of Life Adjusted years [QALYs]) between Baseline and the 12 month visit. The ICER represents the extra costs that have to be incurred for one extra unit of perfect health to be produced. A treatment is determined to be cost-effective if the ICER is below a certain threshold (National Health Systems of European Union have suggested a threshold of 50,000 euros).
Time Frame: 12 months
Population: Cost-utility analysis is based on the 76 participants who completed the study through 12 months.
Measure: Number; unit: Euros
Arm/Group | Adalimumab Treatment
Number analyzed (Participants) | 76
Euros | 13,628

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected in this study with the exception of adverse events leading to withdrawal. Adverse events are collected in the main study NCT 01086033 (GREC-2004-06) and will be reported upon completion of that study.
Description: Only adverse events leading to withdrawal are recorded. Adverse events are collected in the main study NCT 01086033 (GREC-2004-06) and will be reported upon completion of that study. Number of participants at risk (N=124) and adverse event frequency threshold refers only to withdrawals due to adverse event, not overall adverse event reporting.
Arm/Group | Adalimumab Treatment
Serious Adverse Events (participants affected / at risk) | 3/124
Other Adverse Events (participants affected / at risk) | 2/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab Treatment (N=124)
Acute Myocardial Infarction/Coronary Artery Bypass Graft (Cardiac disorders) | 1 — Serious adverse event leading to study withdrawal for one participant. Number of participants at risk (N=124) refers only to study withdrawals due to adverse event, not overall adverse event reporting.
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 — Serious adverse event leading to study withdrawal for one participant. Number of participants at risk (N=124) refers only to study withdrawals due to adverse event, not overall adverse event reporting.
Cellulitis (Skin and subcutaneous tissue disorders) | 1 — Serious adverse event leading to study withdrawal for one participant. Number of participants at risk (N=124) refers only to study withdrawals due to adverse events, not overall adverse event reporting.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab Treatment (N=124)
Rash muculo-papular (Skin and subcutaneous tissue disorders) | 1 — Nonserious adverse event leading to study withdrawal for one participant.Number of participants at risk (N=124) and adverse event reporting frequency threshold refer only to study withdrawals due to adverse event, not overall adverse event reporting.
Hypersensitivity (Immune system disorders) | 1 — Nonserious adverse event leading to study withdrawal in one participant. Number of participants at risk (N=124) and adverse event reporting frequency threshold refer only to study withdrawals due to adverse event, not overall adverse event reporting.

LIMITATIONS AND CAVEATS:
Study NCT 01078116 (P10-159) is a substudy of NCT 01086033(GREC-2004-06). Adverse events were not recorded in this study but will be reported in the main study upon completion. Only adverse events leading to withdrawal are reported in this substudy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.